CLINICAL TRIAL: NCT06091579
Title: A Phase 1, Randomized, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, And Pharmacokinetics of Treprostinil Palmitil Inhalation Powder in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Treprostinil Palmitil Inhalation Powder (TPIP) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INS1009-102
Record Dates: First submitted 2023-10-16; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A (SAD Cohort 1): TPIP (Experimental): Participants in the single ascending dose (SAD) Cohort 1 received a single dose of TPIP at Dose A, Dose B, or Dose C by oral inhalation on Day 1.
  Interventions: Drug: Treprostinil Palmitil Inhalation Powder
- Part A (SAD Cohort 2): TPIP or Placebo (Experimental): Participants in SAD Cohort 2 received a single dose of TPIP at Dose D or matching placebo by oral inhalation on Day 1.
  Interventions: Drug: Treprostinil Palmitil Inhalation Powder; Drug: Placebo
- Part A (SAD Cohort 3): TPIP or Placebo (Experimental): Participants in SAD Cohort 3 received a single dose of TPIP at Dose E or matching placebo by oral inhalation on Day 1.
  Interventions: Drug: Treprostinil Palmitil Inhalation Powder; Drug: Placebo
- Part B (MAD Cohort 1): TPIP or Placebo (Experimental): Participants in the multiple ascending dose (MAD) Cohort 1 received TPIP at Dose B, Dose C or matching placebo, once daily (QD) by oral inhalation on Days 1 through 7.
  Interventions: Drug: Treprostinil Palmitil Inhalation Powder; Drug: Placebo
- Part B (MAD Cohort 2): TPIP or Placebo (Experimental): Participants in MAD Cohort 2 received TPIP up to Dose D or matching placebo, QD by oral inhalation on Days 1 through 7.
  Interventions: Drug: Treprostinil Palmitil Inhalation Powder; Drug: Placebo

INTERVENTIONS:
Drug: Treprostinil Palmitil Inhalation Powder — Oral inhalation using a Plastiape capsule-based dry powder inhaler.
  Other Names: INS1009
Drug: Placebo — Oral placebo inhalation using a Plastiape capsule-based dry powder inhaler.
  Arms: Part A (SAD Cohort 2): TPIP or Placebo; Part A (SAD Cohort 3): TPIP or Placebo; Part B (MAD Cohort 1): TPIP or Placebo; Part B (MAD Cohort 2): TPIP or Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of single and multiple doses of treprostinil palmitil inhalation powder in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* The participant is considered by the investigator to be in good general health as determined by medical history, physical examination findings, vital sign measurements, 12-lead electrocardiogram (ECG) results, and clinical laboratory test results within normal limits or considered not clinically significant by the investigator, at screening.

Exclusion Criteria:

* The participant has an allergy, documented hypersensitivity, or contraindication to the ingredients or to any of the excipients of treprostinil palmitil inhalation powder or treprostinil.
* The participant has used any prescription (excluding hormonal birth control) or over-the-counter medications, including herbal or nutritional supplements, within 14 days before the first dose of study drug and throughout the study.
* The participant has a history of anaphylaxis, previously documented hypersensitivity reaction to any drug.
* The participant has had a surgical procedure that required general anesthesia (or equivalent) within 90 days prior to screening.
* The participant has a body mass index <19.0 or >32.0 kilograms per square meter (kg/m^2) at screening.
* The participant has a history of syncope not due to dehydration or vasovagal syncope (eg, congenital cardiac arrhythmias such as Wolff-Parkinson-White syndrome, nodal tachycardia, ventricular tachycardia, etc).
* The participant has active liver disease or hepatic dysfunction at screening or check-in visits.
* The participant has a history of human immunodeficiency virus (HIV) infection.
* The participant has a history of abnormal bleeding or bruising.
* The participant has a history of malignancy in the past 5 years, with exception of nonmelanoma skin cancer.
* The participant has a current history (within the past 12 months) of substance and/or alcohol abuse.
* The participant is a current user of cigarettes (average of ≥1 cigarette/day) or e-cigarettes within 30 days prior to screening.
* The participant has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at screening or before the first dose of study drug or throughout the study.

Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Parts A and B: Number of Participants who Experienced an Adverse Event (AE) | Up to Day 31 in Part A and Day 37 in Part B
  Safety and tolerability of single and multiple doses of treprostinil inhalation powder will be determined in healthy participants.

SECONDARY OUTCOMES:
Parts A and B: Area Under the Plasma Concentration Versus Time Curve (AUC) of Treprostinil | Part A: Predose and at multiple time points postdose up to Day 4; Part B: Predose and at multiple time points postdose up to Day 10
  Pharmacokinetics of treprostinil following a single and multiple doses will be assessed in healthy participants.
Parts A and B: Area Under the Plasma Concentration Versus Time Curve (AUC) of Treprostinil Palmitil | Part A: Predose and at multiple time points postdose up to Day 4; Part B: Predose and at multiple time points postdose up to Day 10
  Pharmacokinetics of treprostinil palmitil following a single and multiple doses will be assessed in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- USA001, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ismat FA, Usansky HH, Villa R, Zou J, Teper A. Safety, Tolerability, and Pharmacokinetics of Treprostinil Palmitil Inhalation Powder for Pulmonary Hypertension: A Phase 1, Randomized, Double-Blind, Single- and Multiple-Dose Study. Adv Ther. 2022 Nov;39(11):5144-5157. doi: 10.1007/s12325-022-02296-x. Epub 2022 Sep 7. PMID 36070132